CLINICAL TRIAL: NCT02627807
Title: Prospective Non-inferiority Randomized Trial Comparing Clinical Target Volume Based on Disease Extension Risk Atlas and Computer-aided Delineation and Traditional Clinical Target Volume in Radiotherapy for Nasopharyngeal Carcinoma
Brief Title: Clinical Target Volume Based on Disease Extension Risk Atlas and Computer-aided Delineation in Nasopharyngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ying Sun, Chief physician，Deputy director,Assistant dean, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012011
Record Dates: First submitted 2015-12-03; First posted 2015-12-11 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Nasopharyngeal carcinoma; Intensity modulated radiotherapy; Clinical target volume; Clinical trial
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; Induction Chemotherapy; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized CTV (Experimental): Patients receive IMRT using individualized CTV based on disease extension risk atlas and computer-aided delineation. Gemcitabine and cisplatin induction chemotherapy or docetaxel and cisplatin induction chemotherapy and cisplatin 100mg/m² concurrent chemotherapy or cisplatin 80mg/m² concurrent chemotherapy are optional based on clinical classification.
  Interventions: Radiation: IMRT using individualized CTV; Drug: Gemcitabine and cisplatin (induction chemotherapy); Drug: Docetaxel and cisplatin (induction chemotherapy); Drug: Cisplatin 100mg/m² concurrent chemotherapy; Drug: Cisplatin 80mg/m² concurrent chemotherapy
- Traditional CTV (Active Comparator): Patients receive IMRT using traditional CTV. Gemcitabine and cisplatin induction chemotherapy or docetaxel and cisplatin induction chemotherapy and cisplatin 100mg/m² concurrent chemotherapy or cisplatin 80mg/m² concurrent chemotherapy are optional based on clinical classification.
  Interventions: Radiation: IMRT using traditional CTV; Drug: Gemcitabine and cisplatin (induction chemotherapy); Drug: Docetaxel and cisplatin (induction chemotherapy); Drug: Cisplatin 100mg/m² concurrent chemotherapy; Drug: Cisplatin 80mg/m² concurrent chemotherapy

INTERVENTIONS:
Radiation: IMRT using individualized CTV — Intensity modulated radiotherapy (IMRT) using individualized CTV based on disease extension risk atlas and computer-aided delineation is given as 2.13 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 70.29 Gy to the primary tumor.
  Arms: Individualized CTV
Radiation: IMRT using traditional CTV — Intensity modulated radiotherapy(IMRT) using traditional CTV is given as 2.13 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 70.29 Gy to the primary tumor.
  Arms: Traditional CTV
Drug: Gemcitabine and cisplatin (induction chemotherapy) — Induction chemotherapy is optional for patients with T2-4N0-3M0 NPC. Patients who participate in another randomized trial (NCT01872962) at the same time receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 3 cycles before radiotherapy.
  Other Names: Gemcitabine and cisplatin (GP)
Drug: Docetaxel and cisplatin (induction chemotherapy) — Induction chemotherapy is optional for patients with T2-4N0-3M0 NPC. Patients who haven't participated in other trials receive docetaxel (75 mg/m² d1) and cisplatin (75mg/m²,total dose average to d1-d3) every 3 weeks for 3 cycles before radiotherapy.
  Other Names: Docetaxel and cisplatin (TP)
Drug: Cisplatin 100mg/m² concurrent chemotherapy — Cisplatin concurrent chemotherapy is required for patients with T2-4N0-3M0 NPC. Patients who participate another clinical trial (NCT01872962) at the same time receive cisplatin (100mg/m² d1) every 3 weeks for 3 cycles concurrently with radiotherapy.
  Other Names: DDP 100mg/m²
Drug: Cisplatin 80mg/m² concurrent chemotherapy — Cisplatin concurrent chemotherapy is required for patients with T2-4N0-3M0 NPC.Patients who haven't participated in other trials receive cisplatin (80mg/m²,total dose average to d1-d3) every 3 weeks for 3 cycles concurrently with radiotherapy.
  Other Names: DDP 80mg/m²

SUMMARY:
The purpose of this study is to compare individualized clinical target volume (CTV) based on disease extension risk atlas and computer-aided delineation with traditional CTV in intensity modulated radiotherapy (IMRT) for nasopharyngeal carcinoma (NPC), in order to confirm the efficacy and safety.

DETAILED DESCRIPTION:
Patients with non-keratinizing NPC T1-4N0-3M0 (AJCC/UICC staging system 7th edition) are randomly assigned to receive IMRT using individualized clinical target volume (CTV) based on disease extension risk atlas and computer-aided delineation or IMRT using traditional CTV. IMRT is given as 2.13 Gray (Gy) per fraction with five daily fractions per week for 6-7 weeks to a total dose of 70.29 Gy to the primary tumor. Patients with T1N0M0 NPC receive IMRT only. For patients with stage T2-4N0-3M0 NPC, concurrent chemoradiotherapy (CCRT) is required and induction chemotherapy (IC) before CCRT is optional.Patients who participate in another randomized trial (NCT01872962) at the same time receive the protocol chemotherapy. Induction chemotherapy regimens are as follows: gemcitabine (1000 mg/m² d1,8) plus cisplatin (80mg/m² d1) or docetaxel (75mg/m² d1) plus cisplatin (75mg/m², total dose average to d1-d3) every 3 weeks for three cycles. concurrent chemotherapy include cisplatin (100mg/m² d1 or 80mg/m², total dose average to d1-d3) every 3 weeks for three cycles. Our primary endpoint is loco-regional recurrence-free survival (LRRFS) rate. Secondary end points include overall survival (OS) rate, distant metastasis-free survival (DMFS) rate, constituent ratio of local and regional recurrence pattern, toxic effects, quality of life scores and dosimetric parameters of IMRT planning. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type).
* Tumor staged as T1-4N0-3M0 (according to the 7th AJCC edition), based upon the following minimum diagnostic workup within 4 weeks prior to registration:(1) history/physical examination;(2)chest X-ray, PA and lateral OR chest CT OR PET/CT;(3) pre-treatment magnetic resonance imaging (MRI) of nasopharynx and neck, pre-treatment MRI must be done at Sun Yat-sen University Cancer Center;(4) sonography OR CT of upper abdoman OR PET/CT;(5) Bone scan OR PET/CT.
* Satisfactory performance status: Karnofsky scale (KPS) ≥ 70.
* Adequate bone marrow function based upon the complete blood count within 2 weeks prior to registration: leucocyte count ≥ 4000/μL, hemoglobin ≥ 90g/L and platelet count ≥ 100000/μL.
* Adequate hepatic function within 2 weeks prior to registration: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ ULN.
* Adequate renal function within 2 weeks prior to registration: serum creatinine ≤ 133 umol/L or calculated creatinine clearance ≥ 60 ml/min.
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study.
* Patients must be informed of the investigational nature of this study and sign a written informed consent.

Exclusion Criteria:

* Age > 65 or < 18.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer outside head and neck region, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except fine needle aspiration biopsy) to primary tumor or nodes.
* Hearing loss due to sensorineural deafness（except tumor induced conductive hearing loss).
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), emotional disturbance, untreated active infectious disease, and acquired immune deficiency syndrome.
* Prior allergic reaction to the study drugs involved in this protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2015-12; Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Local-regional recurrence-free survival rate | 3-year
  Local-regional recurrence-free survival is calculated from the date of randomization to the date of local or regional recurrence, whichever is first.

SECONDARY OUTCOMES:
Overall survival rate | 3-year
  Overall survival is calculated from the date of randomization to the date of death from any cause.
Distant metastasis-free survival rate | 3-year
  Distant metastasis-free survival is calculated from the date of randomization to the date of the first distant metastasis.
Constituent ratio of local and regional recurrence pattern | 3-year
  Constituent ratio of local and regional recurrence pattern is defined as the proportion of in-field,marginal and out-field recurrence.
Number of participants with adverse events | 3-year
  Incidence of acute and late toxicity
Quality of life score measured by EORTC QLQ-C30 | 3-year
  Quality of life is measured by European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30).
Quality of life score measured by EORTC H&N35 | 3-year
  Quality of life is measured by European Organization for Research and Treatment of Cancer Quality of Life Head and Neck Questionnaire (EORTC QLQ-H&N35).
Target volumes' dose coverage and doses irradiated to organs at risk | 3-year
  For example, relative volume of planning target volume (PTV) receive 110%,95%,93% of the prescription doses;max dose or dose receive by 1% volume of brainstem; et,al.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Sun, Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Lai SZ, Li WF, Chen L, Luo W, Chen YY, Liu LZ, Sun Y, Lin AH, Liu MZ, Ma J. How does intensity-modulated radiotherapy versus conventional two-dimensional radiotherapy influence the treatment results in nasopharyngeal carcinoma patients? Int J Radiat Oncol Biol Phys. 2011 Jul 1;80(3):661-8. doi: 10.1016/j.ijrobp.2010.03.024. Epub 2010 Jul 17. PMID 20643517
- [Background] Lin S, Pan J, Han L, Zhang X, Liao X, Lu JJ. Nasopharyngeal carcinoma treated with reduced-volume intensity-modulated radiation therapy: report on the 3-year outcome of a prospective series. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1071-8. doi: 10.1016/j.ijrobp.2008.12.015. Epub 2009 Apr 11. PMID 19362784
- [Background] Lee N, Xia P, Quivey JM, Sultanem K, Poon I, Akazawa C, Akazawa P, Weinberg V, Fu KK. Intensity-modulated radiotherapy in the treatment of nasopharyngeal carcinoma: an update of the UCSF experience. Int J Radiat Oncol Biol Phys. 2002 May 1;53(1):12-22. doi: 10.1016/s0360-3016(02)02724-4. PMID 12007936
- [Background] Kam MK, Teo PM, Chau RM, Cheung KY, Choi PH, Kwan WH, Leung SF, Zee B, Chan AT. Treatment of nasopharyngeal carcinoma with intensity-modulated radiotherapy: the Hong Kong experience. Int J Radiat Oncol Biol Phys. 2004 Dec 1;60(5):1440-50. doi: 10.1016/j.ijrobp.2004.05.022. PMID 15590175
- [Background] Tham IW, Hee SW, Yeo RM, Salleh PB, Lee J, Tan TW, Fong KW, Chua ET, Wee JT. Treatment of nasopharyngeal carcinoma using intensity-modulated radiotherapy-the national cancer centre singapore experience. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1481-6. doi: 10.1016/j.ijrobp.2009.01.018. Epub 2009 Apr 20. PMID 19386431
- [Background] Hunt MA, Zelefsky MJ, Wolden S, Chui CS, LoSasso T, Rosenzweig K, Chong L, Spirou SV, Fromme L, Lumley M, Amols HA, Ling CC, Leibel SA. Treatment planning and delivery of intensity-modulated radiation therapy for primary nasopharynx cancer. Int J Radiat Oncol Biol Phys. 2001 Mar 1;49(3):623-32. doi: 10.1016/s0360-3016(00)01389-4. PMID 11172942
- [Background] Wolden SL, Chen WC, Pfister DG, Kraus DH, Berry SL, Zelefsky MJ. Intensity-modulated radiation therapy (IMRT) for nasopharynx cancer: update of the Memorial Sloan-Kettering experience. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):57-62. doi: 10.1016/j.ijrobp.2005.03.057. Epub 2005 Jun 2. PMID 15936155
- [Background] Kam MK, Leung SF, Zee B, Chau RM, Suen JJ, Mo F, Lai M, Ho R, Cheung KY, Yu BK, Chiu SK, Choi PH, Teo PM, Kwan WH, Chan AT. Prospective randomized study of intensity-modulated radiotherapy on salivary gland function in early-stage nasopharyngeal carcinoma patients. J Clin Oncol. 2007 Nov 1;25(31):4873-9. doi: 10.1200/JCO.2007.11.5501. PMID 17971582
- [Background] Liang SB, Sun Y, Liu LZ, Chen Y, Chen L, Mao YP, Tang LL, Tian L, Lin AH, Liu MZ, Li L, Ma J. Extension of local disease in nasopharyngeal carcinoma detected by magnetic resonance imaging: improvement of clinical target volume delineation. Int J Radiat Oncol Biol Phys. 2009 Nov 1;75(3):742-50. doi: 10.1016/j.ijrobp.2008.11.053. Epub 2009 Feb 27. PMID 19251378
- [Background] Tang L, Mao Y, Liu L, Liang S, Chen Y, Sun Y, Liao X, Lin A, Liu M, Li L, Ma J. The volume to be irradiated during selective neck irradiation in nasopharyngeal carcinoma: analysis of the spread patterns in lymph nodes by magnetic resonance imaging. Cancer. 2009 Feb 1;115(3):680-8. doi: 10.1002/cncr.24049. PMID 19117352
- [Background] Baujat B, Audry H, Bourhis J, Chan AT, Onat H, Chua DT, Kwong DL, Al-Sarraf M, Chi KH, Hareyama M, Leung SF, Thephamongkhol K, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy in locally advanced nasopharyngeal carcinoma: an individual patient data meta-analysis of eight randomized trials and 1753 patients. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):47-56. doi: 10.1016/j.ijrobp.2005.06.037. PMID 16377415
- [Background] Edge SB, Byrd DR, Compton CC, et al: AJCC Cancer Staging Manual (ed 7th). New York, Springer, 2010
- [Background] Chow SC, Shao J, Wang H: Sample Size Calculations in Clinical Research. New York, Marcel Dekker, 2003
- [Background] Freedman J, Furberg C, DeMets D: Fundamentals of clinical trials. New York, Springer-Verlag, 1998